CLINICAL TRIAL: NCT03701724
Title: Cost-utility Analysis of Maintenance rTMS for Treatment-resistant Depression
Acronym: ACOUSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RC17_0494
Record Dates: First submitted 2018-09-17; First posted 2018-10-10 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Treatment-resistant Depression
Keywords: Major Depressive Disorder; Unipolar depression; Chronic depression; Recurrent depression; Depressive disorder; Magnetic stimulation; Non-invasive brain stimulation; 1 Hertz (Hz) rTMS; Maintenance rTMS; Cost-utility; Efficiency; Medico-economic; Antidepressants
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham rTMS will be used for the arm "without rTMS"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Systematic maintenance rTMS (arm A) (Experimental): Active rTMS treatment followed, for responders, by systematic maintenance rTMS Depression usual medical treatment (psychosocial approach and/or pharmacotherapy and/or, ECT…)
  Interventions: Device: Systematic maintenance rTMS
- rTMS course in case of relapse (arm B) (Experimental): Active rTMS treatment followed, for responders, by additional rTMS courses, in case of relapse Depression usual medical treatment (psychosocial approach and/or pharmacotherapy and/or, ECT…)
  Interventions: Device: rTMS course in case of relapse
- Sham rTMS (arm C) (Sham Comparator): sham rTMS followed, for responders, by either systematic sham mTMS (50%) or additional sham rTMS course in case of relapse(50%) Depression usual medical treatment (psychosocial approach and/or pharmacotherapy and/or, ECT…)
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: Systematic maintenance rTMS — Same parameters as the initial course (session of 8,5 minutes, at 1 Hz, on the right dorsolateral prefrontal cortex (DLPFC) targeting with either neuronavigation or the Beam). The frequency is : 2 sessions / week during 1 month, then 1 session / week during 2 months and finally 1 session every 2 weeks during 8 months.
  Arms: Systematic maintenance rTMS (arm A)
Device: rTMS course in case of relapse — Same parameters as the initial course. The frequency is the same as the initial course: one daily session on 5 consecutive working days from Monday to Friday for at least 20 to 30 sessions over 4 to 6 weeks.
  Arms: rTMS course in case of relapse (arm B)
Device: sham rTMS — The sham stimulation consists of the identical rTMS procedure at the identical location using a commercial figure-eight sham coil. However, it does not produce the identical tactile sensation. A local electrical stimulation will be delivered with two disposable Electromyogram (EMG) electrodes using a transcutaneous electrical nerve stimulation (TENS) Stimulator.
  Arms: Sham rTMS (arm C)

SUMMARY:
Treatment resistant depression (TRD) is a frequent, debilitating condition mostly treated by antidepressants. Repeated magnetic transcranial stimulation (rTMS) has proven adjuvant efficacy in TRD in the acute phase of treatment with a very good tolerance and acceptability. Maintenance rTMS (mTMS) is a strategy consisting in adding regular single TMS sessions after response to an acute course in order to keep the benefit of initial treatment over several month or years. Demonstrating that rTMS is efficient to improve long-term prognosis and decrease economic burden would have a tremendous impact in clinical practice in psychiatry. Thus the investigator's aim is to analyze the long term impact of mTMS treatment on costs, but also quality of life and clinical issues.

DETAILED DESCRIPTION:
TRD is associated with enormous social, economic, and personal costs. In literature, psychosocial and pharmacological interventions showed limited one year long-term efficacy in terms of relapse (only 10% of sustained remission at one-year follow-up actually) and quality of life due to refractoriness, observance and adverse effects. In the recent years the field of non-invasive brain stimulation became more mature with an increasing level of evidence reaching Level 1 for rTMS as curative treatment for depression in international guidelines. It is a safe and well tolerated treatment but with still high relapse rate at 6 month and one year (comparable to those former described for ECT). mTMS is a promising tool (as it was proven for ECT) to achieve sustained response several month after treatment in a significant proportion of patients. Little is known about its long-term economic and social benefit which is a crucial question given its time consuming nature. To date there is no large Randomized Clinical Trial (RCT) assessing the long-term health economic interest or adjuvant mTMS compared to treatment as usual (TAU) alone in unipolar TRD . This study is a double-blind randomized controlled trial aiming at determining a 12 month cost-utility analysis, according to collective perspective, of two different modalities of rTMS (systematic mTMS or curative rTMS in case of relapse) for TRD compared to TAU alone. The secondary aims are to describe 24 month cost-utility, longitudinal clinical issues in terms of mood and quality of life, prognosis factors, as well as TAU actual strategies in that population.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 MADRS >19
* Episode duration: 12 weeks to 3 years.
* 2 to 4 unsuccessful treatment lines (including antidepressants, and potentialization agents lithium and quetiapine) despite adequate dosage and duration (6 weeks stable posology)
* Ability to consent and express informed consent, to answer questionnaires and to go to follow-up visits.
* Affiliation to social security

Exclusion Criteria:

* Bipolar disorder
* Schizophrenia and other psychotic disorders
* Mental retardation or developmental disorder
* Substance abuse or dependence
* Depression symptoms better explained by medical conditions
* Neurologic conditions (e.g.,previous epilepsy or unexplained seizures, stroke, trauma, infection, metabolic disease, severe migraines, multiple sclerosis, brain tumor)
* Presence of at least one contra-indication to rTMS
* Pregnancy/breast-feeding
* Patient who previously received 5 lines or more pharmacological treatment for the current episode (excluding symptomatic psychotropic drugs, e.g. benzodiazepines and hypnotics)
* Former use of electroconvulsive therapy or rTMS within the current episode.
* Previous failure of adequate ECT (at least 12 well conducted sessions) or rTMS course (at least 20 well conducted sessions) in the medical history.
* History of at least two courses of ECT, previous need for maintenance ECT.
* Protection measure : maintenance of justice, tutelage, legal guardianship
* Woman of childbearing age without effective contraception
* Liberty deprivation (e.g. incarceration, therapeutic injunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cost-utility ratio, according to collective perspective of rTMS use in TRD compared to conventional therapeutic approaches without active rTMS. | 12 months
  The utility will be measured by :
  Quality Adjusted Life Year (QALYs) as estimated from responses to the Euroqol-5 Dimensions (EQ-5D) health-related quality of life questionnaire. The questionnaire focuses on 5 dimensions: mobility, personal autonomy, current activities, pain/discomfort and anxiety/depression. For each of these dimensions, 3 answers are possible.
  The costs will be measured by the addition of the following costs:
  Drugs dispensing via Health insurance database "National system of information of the French health insurance" (SNIIRAM), hospitalizations, work stoppages and care consumption collected in a declarative patient questionnaire.

SECONDARY OUTCOMES:
Cost-utility ratio, according to collective perspective of rTMS use in TRD compared to conventional therapeutic approaches without active rTMS. | 24 months
  Quality Adjusted Life Year (QALYs) as estimated from responses to the Euroqol-5 Dimensions (EQ-5D) health-related quality of life questionnaire
  The costs will be measured by the additional of the following costs:
  Drugs dispensing via Health insurance database SNIIRAM, hospitalizations, work stoppages and care consumption collected in a declarative patient questionnaire
Budget impact analysis of spreading the most efficient strategy for using rTMS (systematic mTMS or rTMS course in case of relapse). | 5 years
  Comparison of intervention costs on the study sample and projection of these costs over 5 years, from the health insurance and hospital perspectives
Major depressive disorder history | Baseline
  This outcome will be assessed by patient interview, with the following data (not exhaustive): date of initial symptoms, length of the current episode, family antecedents of mood disorders.
Level of depression treatment-resistance | Baseline
  Maudsley Staging model score: a multidimensional tool to quantify treatment resistance in depression. It evaluates 5 dimensions: 1) length of the current depressive episode, 2) symptomatic intensity, 3) failure of the antidepressant drugs, 4) Increase treatment 5) use of Electro-convulsive therapy. The total score ranges from 3 to 15. 15 being the highest level of treatment resistance.
professional status | Baseline,12 months and 24 months
  patient's professional status (active, unemployed, retired...)
marital status | Baseline,12 months and 24 months
  patient's marital status (married, widow, single...)
Response rate | 12 months and 24 months
  Response is defined as follows: decrease of the MADRS score by at least 50% compared to baseline score. MADRS stands for Montgomery-Asberg Depression Rating Scale. It is used to measure the severity of depressive episodes in patients with mood disorders. The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. A score from 0 to 6 being normal/symptom absent and a score >34 being severe depression.
Remission rate | 12 months and 24 months
  Remission is defined as follows: MADRS score ≤ 10 (see detailed description of MADRS in outcome 8)
Relapse-free survival | 12 months and 24 months
  Number of patients with no relapse. Relapse is defined as follows: MADRS ≥ 20 (see detailed description of MADRS in outcome 8)
MADRS score | Baseline, 2 months, 6 months , 9 months, 12 months, 18 months, 24 months
  MADRS score (see detailed description of MADRS in outcome 8)
Beck Depression Inventory (BDI) score | Baseline, 2 months, 6 months , 9 months, 12 months, 18 months, 24 months
  The BDI is 13-item multiple-choice self-report inventory, for measuring the severity of depression. The global score is an addition of each item's score and ranges from 0 (minimal depression) to 39 (severe depression).
Clinical Global Impression (CGI) score | Baseline, 2 months, 6 months , 9 months, 12 months, 18 months, 24 months
  The Clinical Global Impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. Each scale is rated from 0 to 7. 0 being the best level and 7 the worst level.
Adverse events linked to the medical treatment for depression | 24 months
  Number and types of adverse events linked to the medical treatment for depression
Declarative drug compliance via the MARS (Medication Adherence Report Scale) | baseline, 12 months and 24 months
  MARS is the Medication Adherence Report Scale, including 10 questions, the global score ranges from 0 to 10, 0 corresponds to the worst drug compliance and 10 to an excellent drug compliance
Declarative drug compliance via the CRS (Clinician Rating Scale) | baseline, 12 months and 24 months
  CRS is the Clinician Rating Scale , including 7 questions, the global score ranges from 1 to 7, 7 being the worst level of drug compliance.
Treatment(s) switch(es) | Baseline, 2 months, 6 months , 9 months, 12 months, 18 months, 24 months
  Number of treatment switches per patient
Treatment(s) dose increase | Baseline, 2 months, 6 months , 9 months, 12 months, 18 months, 24 months
  Number of drug(s) dose(s) increases prescribed to the patient
Treatments combination(s) | Baseline, 2 months, 6 months , 9 months, 12 months, 18 months, 24 months
  List of drugs (name) prescribed to the patient
Rate of suicide attempts and suicides | 12 months and 24 months
  number of suicide attempts and suicides per patient
Patient's quality of life | baseline,12 months and 24 months
  Short-Form 36 (SF 36) questionnaire: instrument used to assess multidimensional health-related quality of life, which measures 8 health related parameters: physical function, social function, physical role, emotional role, mental health, energy, pain, general health perceptions
Response rate at the end of rTMS courses | 1 month after each rTMS treatments
  Response is defined as follows: decrease of the MADRS score by at least 50% compared to baseline score (see detailed description of MADRS in outcome 8)
Remission rate at the end of rTMS courses | 1 month after each rTMS treatments
  Remission is defined as follows: MADRS score ≤ 10 (see detailed description of MADRS in outcome 8)
Number of days between the successive rTMS courses | 24 months
  Number of days between end of rTMS course X and beginning of course X+1, for each patient
Total number of rTMS sessions | 24 months
  total number of rTMS sessions per patient
Time between relapses | 24 months
  Number of days between relapses, per patient
Compliance with rTMS | 24 months
  number of missed sessions over the number of planned sessions, per patient
Patient acceptability of the rTMS technique: Analog Visual Scale | 24 months
  Analog Visual Scale of acceptability of the rTMS completed by the patient, ranging from 0 to 10. 0 being "not acceptable" and 10 being "totally acceptable"

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Bulteau, MD, Principal Investigator — Nantes University Hospital
Locations (19):
- France (19):
  - CHU d'Angers, Angers
  - CHRU de Besançon, Besançon
  - CH le Vinatier Lyon, Bron
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - Clinique de Vontes, Esvre-sur-Indre
  - EPSM de Lille, Lille
  - CH Esquirol - Limoges, Limoges
  - CHU de Montpellier, Montpellier
  - Nantes University Hospital, Nantes
  - EPS de Ville-Evrard, Neuilly-sur-Marne
  - GH PItié Salpétrière, Paris
  - GHU Psychiatrie Ste Anne, Paris
  - CH Henri Laborit (Poitiers), Poitiers
  - Centre hospitalier Guillaume Regnier Rennes, Rennes
  - CH du Rouvray - Rouen, Rouen
  - CHU de Toulouse, Toulouse
  - CHU de Tours / CHRU de Tours, Tours

REFERENCES:
- [Derived] Bulteau S, Laurin A, Volteau C, Dert C, Lagalice L, Schirr-Bonnans S, Bukowski N, Guitteny M, Simons L, Cabelguen C, Pichot A, Tessier F, Bonnin A, Lepage A; ACOUSTIM Investigators Group; HUGOPSY Network; Vanelle JM, Sauvaget A, Riche VP. Cost-utility analysis of curative and maintenance repetitive transcranial magnetic stimulation (rTMS) for treatment-resistant unipolar depression: a randomized controlled trial protocol. Trials. 2020 Apr 5;21(1):312. doi: 10.1186/s13063-020-04255-9. PMID 32248820